CLINICAL TRIAL: NCT03791203
Title: A Randomized Controlled Trial on the Effectiveness and Adherence of Modified Alternate-day Calorie Restriction (MACR) in Improving Activity of Non-Alcoholic Fatty Liver Disease
Brief Title: Effectiveness and Adherence of Modified Alternate-day Calorie Restriction (MACR) in Non-Alcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Muhammad Izzad Bin Johari, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 304/PPSP/61313173
Record Dates: First submitted 2018-12-16; First posted 2019-01-02 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Non-alcoholic fatty liver disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Participants who fulfilled the selection criteria were randomly assigned to the modified alternate-day calorie restriction (MACR) group or the control group after a 2 week run-in period. During the 2 weeks, participants were required to keep their body weight stable by maintaining their usual eating habits and their daily activities. Randomization was performed using a random number generator with recruitment aimed for three MACR participants for every control participant by principal investigator.
Who Masked: Participant
Masking Description: Participants were blinded after assignment to interventions or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calorie restriction (MACR) (Experimental): Participants restricted 70% of their energy needs over 24 hours on a calorie restriction day alternate with a feeding day for the next 24 hours, where they were allowed eating (ad libitum). The calorie restriction and feeding days begun at 9 am each day, and on the calorie restriction day, meals were consumed between 2 pm and 8 pm to ensure that they underwent the same duration of calorie restriction. On each calorie restriction day, they were allowed energy-free beverages and sugar-free gum and encouraged to drink plenty of water. Diet plans were self-selected using detailed individualized food portion lists, meal plans, and recipes. Participants received phone calls from the investigator and four 2-weekly appointments with a dietitian. Adverse experiences were assessed every 2 weeks.
  Interventions: Behavioral: Calorie restriction (MACR)
- Control group (No Intervention): Participants in the control group continued their usual habitual diet for 8 weeks. No specific dietary advice or educations were provided throughout the entire trial.

INTERVENTIONS:
Behavioral: Calorie restriction (MACR) — This was a randomized, single-blind controlled trial with modified alternate-day calorie restriction (MACR) as the active intervention and normal habitual diet as control at Hospital University of Sains Malaysia.
  Other Names: Modified Alternate-day Calorie Restriction (MACR)
  Arms: Calorie restriction (MACR)

SUMMARY:
There is no effective therapy for non-alcoholic fatty liver disease (NAFLD), although intensive calorie restriction is typically recommended but dietary adherence is an issue. Currently, there are no studies had been focusing the effect of Modified Alternate Day Calorie Restriction in NAFLD patient focusing on changes in liver steatosis and fibrosis.

DETAILED DESCRIPTION:
Disease activity and progression of non-alcoholic fatty liver disease (NAFLD) to non-alcoholic steatohepatitis (NASH) and cirrhosis can be highly variable, where 2-3% will eventually progress to end-stage liver diseases. With the rising prevalence of metabolic syndrome and obesity, NAFLD has become the most frequent form of chronic liver disease in the West but also in Asia.

There are good evidence that weight loss is effective in improving liver histology in NAFLD, for example, 31 obese patients with NASH was randomised into intensive lifestyle changes over 48 weeks versus structured basic education only, and the intensive lifestyle group showed significant improvements in steatosis, necrosis, and inflammation. Intense calorie restriction is the recommended form of dietary strategy for management of NAFLD. Even though such intense dietary strategy has proven to be effective, some patients find it difficult to adhere and maintain.

On the other hand, intermittent fasting achieves more consistent weight loss by improving adherence, as intermittent fasting only requires calorie restriction every other day compared to conventional form of daily calorie restriction. Alternate day calorie restriction can be divided into two components, a 'feed day' and a 'fast day' where food is consumed ad libitum for 24 hours period alternating with either complete or partial (modified) calorie restriction for the next 24 hours. MACR, the dietary strategy employed in the investigator's study, restricts 70% of an individual's daily requirement of calorie per day. There are other forms of intermittent fasting, for example, 2-4 days of ad libitum feeding alternating with 2-4 days of calorie restriction.

Currently, there are no approved pharmacological therapies for NAFLD, and many guidelines advocate recommendation with a focus on controlling risk factors and lifestyle interventions that include dietary and physical activities. No specific NAFLD trials have evaluated the effectiveness of modified form of intermittent fasting in the control of NAFLD activity.

ELIGIBILITY:
Inclusion Criteria:

* Have elevated ALT or AST level (ALT >41 or AST>34 IU/L)
* No evidence of other forms of liver diseases
* For those with diabetes mellitus and dyslipidaemia, they must be on a stable therapy for at least 6 months prior to study enrolment

Exclusion Criteria:

* Significant alcohol consumption (> 1 standard drink per day)
* Pregnancy
* Involvement in an active weight loss program or taking weight loss medications
* Substance abuse and significant psychiatric problems.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline shear wave elastography (SWE) at 8 weeks | Change from baseline at 8-week
  Through the intercostal approach, SWE measurements were performed in the right liver lobe, at the supine position with the right arm in maximal abduction. The sonographer, assisted by an ultrasonic time-motion image, located a liver portion of at least 6 cm thick, free of large vascular structures. Once the measurement area had been located, the sonographer pressed the probe button to start an acquisition. Patients were asked to hold their breath for about five seconds, while the stiffness of the region of interest was measured and 10 measurements were made for each patient and the median average value of those measurements was recorded in kilopascals (kPa: metric).
Change from baseline liver steatosis at 8 weeks | Change from baseline at 8-week
  Ultra-sonographic measurements including liver steatosis and shear wave elastography (SWE) were performed with the SuperSonic Imagine's Aixplorer® Ultrasound machine (Super Sonic Image, Aix-en Provence, France). All measurements were performed by a single sonographer where the inter-observer agreement level with another experienced sonographer was 85%.
Concentration of high-density lipoprotein (HDL) | Change from baseline at 8-week
  Blood samples (8-10 hours of fasting blood samples) were collected from participants at 8-10 am at baseline and 8-week post intervention for biochemical analysis. It was measured in mmol/L.
Concentration of low-density lipoprotein (LDL) | Change from baseline at 8-week
  Blood samples (8-10 hours of fasting blood samples) were collected at 8-10 am at baseline and 8-week post intervention for biochemical analysis. It was measured in mmol/L.
Concentration of triglycerides (TG) | Change from baseline at 8-week
  Blood samples (8-10 hours of fasting blood samples) were collected at 8-10 am at baseline and 8-week post intervention for biochemical analysis. It was measured in mmol/L.
Concentration of total cholesterol (TC) | Change from baseline at 8-week
  Blood samples (8-10 hours of fasting blood samples) were collected at 8-10 am at baseline and 8-week post intervention for biochemical analysis. It was measured in mmol/L.
Concentration of fasting blood sugar (FBS) | Change from baseline at 8-week
  Blood samples (8-10 hours of fasting blood samples) were collected at 8-10 am at baseline and 8-week post intervention for biochemical analysis. It was measured in mmol/L.
Concentration of alanine aminotransferase (ALT) | Change from baseline at 8-week
  Blood samples (8-10 hours of fasting blood samples) were collected at 8-10 am at baseline and 8-week post intervention for biochemical analysis. It was measured in U/L.
Concentration of aspartate aminotransferase (AST) | Change from baseline at 8-week
  Blood samples (8-10 hours of fasting blood samples) were collected at 8-10 am at baseline and 8-week post intervention for biochemical analysis. It was measured in U/L.

SECONDARY OUTCOMES:
Dietary plan adherence | At 8-week
  Adherence data were assessed each week as percentage of adherence

CONTACTS AND LOCATIONS:
Overall Officials: Yeong Yeh Lee, MD, PhD, Principal Investigator — Universiti Sains Malaysia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-08-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT03791203/Prot_SAP_000.pdf
  • Informed Consent Form (2015-10-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT03791203/ICF_001.pdf